CLINICAL TRIAL: NCT04895267
Title: Low-field Thoracic Magnetic Stimulation Increases Peripheral Oxygen Saturation Levels in Coronavirus Disease (COVID-19) Patients: a Single-blind, Sham-controlled, Crossover Study
Brief Title: Low-field Thoracic Magnetic Stimulation Increases Peripheral Oxygen Saturation Levels in COVID-19 Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Elias Manjarrez (Other)
Collaborators: National Council of Science and Technology, Mexico (Other)
Responsible Party: Sponsor-Investigator, Elias Manjarrez, Profesor Investigador Titular, Hospital Univeristario Benemerita Universidad Autonoma de Puebla
Organization: Hospital Univeristario Benemerita Universidad Autonoma de Puebla (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Registration number: 818
Record Dates: First submitted 2021-05-15; First posted 2021-05-20 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: COVID-19; Acute Respiratory Failure; Oxygen Deficiency
Keywords: SpO2; low-field thoracic magnetic stimulation; SARS-CoV-2
MeSH Terms: conditions — COVID-19; Hypoxia

STUDY DESIGN:
Intervention Model Description: Arms:
  The investigators designed a single-blind, sham-controlled, crossover study on COVID-19 participants who underwent two sessions of the study (real and sham Low-field thoracic magnetic stimulation, LF-ThMS), and other COVID-19 participants who underwent only the real LF-ThMS.
  Sham comparator:
  For sham exposure, the coils were positioned in the same coordinates in the same COVID-19 participants, but the LF-ThMS pulse generator was not turned on.
Who Masked: Participant, Care Provider
Masking Description: The investigators designed a single-blind, sham-controlled, crossover study, in which the COVID-19 participants were blinded for the real LF-ThMS or sham stimulation conditions.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real Low-field thoracic magnetic stimulation (LF-ThMS) (Experimental): Crossover, single-blind session of low field thoracic magnetic stimulation (real LF-ThMS)
  Interventions: Device: Low-field thoracic magnetic stimulation (LF-ThMS)
- Sham Low-field thoracic magnetic stimulation (LF-ThMS) (Sham Comparator): In the same patients the coils are positioned in the same coordinates for sham exposure, but the pulse generator is not turned on. Subjects are blinded for the real LF-ThMS or sham stimulation conditions.
  Interventions: Device: Low-field thoracic magnetic stimulation (LF-ThMS)

INTERVENTIONS:
Device: Low-field thoracic magnetic stimulation (LF-ThMS) — A 30 minutes session of low-field thoracic magnetic stimulation (LF-ThMS) is planned for each participant.

SUMMARY:
This study aimed to present a proof-of-concept that a 30 minutes single-session of low-field thoracic magnetic stimulation (LF-ThMS) on the dorsal thorax can be employed to increase oxygen saturation (SpO2) levels in coronavirus disease (COVID-19) participants significantly. The investigators (Saul M. Dominguez-Nicolas and Elias Manjarrez) hypothesized that the variables associated with LF-ThMS, as hyperthermia, frequency, and magnetic flux density in the dorsal thorax, might be correlated to SpO2 levels in these participants. The investigators designed a single-blind, sham-controlled, crossover study on COVID-19 participants who underwent two sessions of the study (real and sham LF-ThMS), and other COVID-19 participants who underwent only the real LF-ThMS.

DETAILED DESCRIPTION:
The severe acute respiratory syndrome coronavirus (CoV)-2 (SARS-CoV-2) may cause low SpO2 and respiratory failure in COVID-19 patients. Hence the increase of SpO2 levels could be crucial for the quality of life and recovery of these patients. In this clinical trial, the investigators (Saul M. Dominguez-Nicolas and Elias Manjarrez) propose that an electromagnetic device termed low-field thoracic magnetic stimulation (LF-ThMS) system could be employed for 30 minutes to increase SpO2 levels in COVID-19 participants. This device non-invasively delivers a pulsed magnetic field from 100 to 118 Hz and 10.5 to 13.1 milliTesla (mT) (i.e., 105 to 131 Gauss) to the dorsal thorax. In line with preliminary studies, the scientific literature, and other devices currently used in musculoskeletal magnetic therapy, these frequencies and magnetic flux densities are safe for the participants. The investigators designed a single-blind, sham-controlled, crossover study on COVID-19 participants who underwent two sessions of the study (real and sham LF-ThMS) and other participants who underwent only the real LF-ThMS. The study design includes a 30 minutes single-session of LF-ThMS to avoid confounding factors related to the spontaneous recovery by natural immunity, common in many COVID-19 patients several days after the contagion. Here the LF-ThMS protocol is not intended to demonstrate its use as therapy but is instead designed to examine the following physiological hypothesis. The hypothesis that there is a statistically significant correlation between magnetic flux density, frequency, or temperature associated with the real LF-ThMS and SpO2 levels in COVID-19 participants. In this context, the present clinical trial is relevant because it could motivate future randomized clinical trials to examine whether the LF-ThMS could be helpful as a potential therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants diagnosed with mild to moderate COVID-19 disease without pneumonia.
* COVID-19 participants with a SpO2 level less or equal to 90 %, exhibiting difficulty breathing, but not intubated.
* COVID-19 participants with similar pharmacological treatment against COVID-19.
* 20-85 years old

Exclusion Criteria:

* COVID-19 patients with acute respiratory failure requiring urgent intubation
* COVID-19 patients with impaired consciousness
* Pregnant woman
* Patients with metallic implants in the thorax, abdomen, or arms, or with electronic medical devices such as pacemakers
* Children

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2020-07-03 (Actual); Primary Completion 2022-08-03 (Estimated); Study Completion 2022-09-17 (Estimated)

PRIMARY OUTCOMES:
1. Change from Baseline Peripheral Oxygen Saturation levels (SpO2) during the intervention | 30 minutes
  1. Change from Baseline Peripheral Oxygen Saturation levels (SpO2) at 30 minutes of LF-ThMS intervention.
2. Peripheral Oxygen Saturation levels (SpO2) after the intervention | 6 months
  2. To evaluate the safety of the intervention, SpO2 levels also are evaluated up to 6 months after the 30 minutes single session of LF-ThMS intervention.

SECONDARY OUTCOMES:
1. Magnetic hyperthermia | 30 minutes
  Coils temperature on the dorsal thorax is measured every 5 minutes during a 30 minutes LF-ThMS session (sham and real).
2. Frequency of the pulsed magnetic stimulation | 30 minutes
  The frequency of the pulsed LF-ThMS on the dorsal thorax is measured every 5 minutes during a 30 minutes LF-ThMS session (sham and real).
3. Magnetic flux density of the pulsed magnetic stimulation | 30 minutes
  The magnetic flux density of the pulsed LF-ThMS on the dorsal thorax is measured every 5 minutes during a 30 minutes LF-ThMS session (sham and real).

CONTACTS AND LOCATIONS:
Overall Officials: Elias Manjarrez, PhD, Principal Investigator — Benemérita Universidad Autónoma de Puebla; Saul M Dominguez-Nicolas, PhD, Principal Investigator — Universidad Veracruzana
Locations (1):
- Benemérita Universidad Autónoma de Puebla, Puebla City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
The investigators (Saul M. Dominguez-Nicolas and Elias Manjarrez) plan to make individual participant data (IPD) collected in this study.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starting 6 months after publication
Access Criteria: open access

REFERENCES:
- [Derived] Dominguez-Nicolas SM, Manjarrez E. Low-field thoracic magnetic stimulation increases peripheral oxygen saturation levels in coronavirus disease (COVID-19) patients: A single-blind, sham-controlled, crossover study. Medicine (Baltimore). 2021 Oct 8;100(40):e27444. doi: 10.1097/MD.0000000000027444. PMID 34622862